CLINICAL TRIAL: NCT06590285
Title: Diagnostic Refinement and Educational Approaches in Managing Bone Marrow Transplantation (DREAM-BMT)
Brief Title: Diagnostic Refinement and Educational Approaches in Managing Bone Marrow Transplantation
Acronym: DREAM-BMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Health (Other)
Collaborators: Scripps Clinic (Other)
Responsible Party: Principal Investigator, Jacob New, Principal Investigator, Scripps Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-24-8378
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: GVHD; Bone Marrow Transplant Complications

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to standard of care monitoring or an educational intervention aimed at improving sleep and activity management during the transplantation process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Monitoring (No Intervention): Usual care will be undergoing alloHSCT without any additional sleep-related educational interventions.
- App-based Educational Intervention (Experimental): The intervention is a pioneering, evidence-based educational program designed to optimize sleep and physical activity outcomes in patients undergoing allogeneic Hematopoietic Stem Cell Transplantation (alloHSCT).
  Interventions: Behavioral: App-based Educational Intervention

INTERVENTIONS:
Behavioral: App-based Educational Intervention — The program's educational content is designed to engage patients in the science of sleep and recovery. Segments like "The Sleep Adventure" demystify complex neurobiological processes in an accessible format, aligning with emerging trends in patient education that focus on engagement and knowledge empowerment. Concurrently, the program's physical activity component is meticulously crafted, offering safe, supportive exercises that correspond with the treatment stages of alloHSCT patients. This aspect draws upon evidence highlighting the importance of sustained physical activity during intensive treatments to enhance overall recovery and quality of life. Additionally, the program comprehensively addresses sleep disturbances, prevalent in HSCT patients, through in-depth exploration and evidence-based, non-pharmacologic management strategies, reflecting the significant impact of sleep quality on patient recovery and long-term health outcomes.
  Arms: App-based Educational Intervention

SUMMARY:
This randomized, phase I/II, open-label study will investigate the efficacy and safety of an educational sleep intervention vs standard of care in adults undergoing alloHSCT. The randomization target in this pilot phase is 60 patients.

DETAILED DESCRIPTION:
To facilitate rapid randomization and baseline collection of patient samples in the patient's home environment, screening activities and assessment of inclusion and exclusion criteria will begin once the patient is identified as transplant eligible at the bone marrow transplant meeting. The patient will subsequently be contacted by a study investigator to explain the study, including its potential benefits and risks.

Patients meeting all inclusion and exclusion criteria will be randomized 1:1 to receive either educational intervention or standard of care therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 or older at the time of study informed consent.
* Have plan to undergo alloHSCT from any donor source using bone marrow, peripheral blood stem cells, or cord blood. Recipients of non-myeloablative, myeloablative and reduced intensity conditioning are eligible.
* Patients have access to digital device capable of downloading study app
* Patients able to read study documents and able to complete informed consent within the study app

Exclusion Criteria:

* Failed prior alloHSCT within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2031-03-01 (Estimated); Study Completion 2033-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective Sleep Measurement | Continuous measurement throughout the study duration (from 2 weeks prior to alloHSCT to 100 days post-alloHSCT)
  A wearable device will continuously measure objective sleep quality. The outcome will be reported as the average sleep duration (in minutes per day) over the study period. Data will be aggregated for the entire duration of the study.

SECONDARY OUTCOMES:
Objective activity measurement | Continuous measurement throughout the study duration (from 2 weeks prior to alloHSCT to 100 days post-alloHSCT).
  A wearable device will continuously measure physical activity. The outcome will be reported as the average activity duration (in minutes per day) over the study period.
Subjective sleep quality | Measurements will occur 12 days prior to alloHSCT, 10 days after alloHSCT and 60 days after alloHSCT
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), with measurements taken at 12 days prior to hospitalization for alloHSCT, 10 days after alloHSCT, and 60 days after alloHSCT. The PSQI is a validated questionnaire that includes a combination of Likert-type and open-ended questions, which are converted to scaled scores following the PSQI guidelines. Respondents indicate the frequency of specific sleep difficulties over the past month and rate their overall sleep quality. Scores for each component range from 0 to 3. Scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.

OTHER OUTCOMES:
Incidence of acute GVHD | Monitoring will occur from day of alloHSCT to 100 days post alloHSCT.
  The incidence of acute GVHD will be evaluated through clinical assessment by the treating physician. The outcome will be reported as the number of days from alloHSCT to the onset of acute GVHD.

CONTACTS AND LOCATIONS:
Overall Officials: Jake New, MD, PhD, Principal Investigator — Scripps Clinic
Locations (1):
- Scripps Health, San Diego, California, United States